CLINICAL TRIAL: NCT00103428
Title: A Phase 1/2a Dose-Escalation Trial of Intravenous CG7870 in Combination With Docetaxel in Chemotherapy-Naïve Patients With Metastatic Hormone-Refractory Prostate Cancer
Brief Title: Intravenous CG7870 in Combination With Docetaxel in Patients With Metastatic Hormone-Refractory Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V-0039
Record Dates: First submitted 2005-02-08; First posted 2005-02-09 (Estimated); Last update posted 2006-02-02 (Estimated); Status verified 2006-01

CONDITIONS: Prostate Cancer
Keywords: chemotherapy; prostate cancer; cancer; metastatic; hormone refractory; chemotherapy naive; dose escalation
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Biological: CG7870

SUMMARY:
V-0039 is a Phase 1/2 dose escalation trial of CG7870 in combination with Docetaxel in metastatic hormone-refractory patients who have not received chemotherapy.

All patients will receive docetaxel. In the dose escalation phase of the study, patients will receive treatment intravenously with CG7870 at one of up to four dose levels. In the Phase 2 portion of this study, additional patients will be added at the maximum tolerated dose that is determined in Phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Metastatic prostate cancer deemed to be unresponsive or refractory to hormone therapy (after discontinuation of anti-androgen therapy)
* Detectable metastases by bone scan, and/or CT scan, and/or MRI, and/or CXR
* ECOG performance status 0-1

Exclusion Criteria:

* Transitional cell, small cell, neuroendocrine, or squamous cell prostate cancer
* History of deep vein thrombosis or pulmonary embolus
* Patients taking anticoagulants (such as coumadin or Heparin). The use of aspirin while on study is acceptable.
* History of a bleeding disorder or recent clinically significant bleeding
* Seropositive for HIV
* History of Hepatitis B, Hepatitis C, or chronic liver disease
* Prior gene therapy or immunotherapy
* Prior chemotherapy for prostate cancer
* Radiation therapy within 4 weeks of the first treatment.
* History of myocardial infarction within 6 months of the first treatment
* History of cerebrovascular accident
* History of previous malignancy, except for the following: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, adequately treated Stage I or II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 5 years
* Evidence of active prostatitis
* Known hypersensitivity to docetaxel or to other drugs formulated with polysorbate 80

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69
Dates: Start 2004-08

PRIMARY OUTCOMES:
Metastatic hormone refractory prostate cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Crowley Medical Research Center, Dallas, Texas, United States